CLINICAL TRIAL: NCT06509321
Title: Comparative Study Between Loupe-Assisted Varicocelectomy With Nitroglycerin Instillation Versus Microscopic Varicocelectomy
Brief Title: Comparison Between Loupe-Assisted Varicocelectomy With Nitroglycerin Instillation and Microscopic Varicocelectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fayoum University Hospital (Other)
Responsible Party: Principal Investigator, Khaled Mohyelden, Professor of urology, Fayoum University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: M 652
Record Dates: First submitted 2024-06-02; First posted 2024-07-19 (Actual); Last update posted 2024-07-23 (Actual); Status verified 2024-07

CONDITIONS: Varicocele
MeSH Terms: conditions — Varicocele

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- subinguinal loupe-assisted varicocelectomy (LV) (Active Comparator): we are using nitroglycerine instillation during loupe assisted varicocelectomy to enhance its efficacy by the vasodilatation effect of Nitroglycerine
  Interventions: Procedure: subinguinal loupe-assisted varicocelectomy (LV)
- subinguinal microscopic varicocelectomy (MV) (Active Comparator): we are using surgical microscope to perform varicocelectomy as control group
  Interventions: Procedure: subinguinal microscopic varicocelectomy (MV)

INTERVENTIONS:
Procedure: subinguinal loupe-assisted varicocelectomy (LV) — to assess the efficacy and safety of sub inguinal loupe-assisted varicocelectomy with nitroglycerin instillation as a vasodilator and compare its results versus subinguinal microscopic varicocelectomy
  Arms: subinguinal loupe-assisted varicocelectomy (LV)
Procedure: subinguinal microscopic varicocelectomy (MV) — we are using surgical microscope to perform varicocelectomy as control group
  Arms: subinguinal microscopic varicocelectomy (MV)

SUMMARY:
This study aims to compare the efficacy and safety of sub inguinal loupe-assisted varicocelectomy with nitroglycerin instillation as a vasodilator and compare it versus sub inguinal microscopic varicocelectomy

DETAILED DESCRIPTION:
This study will include 60 patients with clinical varicocele indicated for varicocelectomy admitted to the Urology Department, at Fayoum University Hospital. The patients will be prospectively randomized into two groups (with ratio 1:1, 30 patients for each group).

* Group A will be treated with subinguinal loupe-assisted varicocelectomy (LV) technique with nitroglycerin instillation as a vasodilator.
* Group B will be treated with subinguinal microscopic varicocelectomy (MV) technique.

Informed consent will be obtained from all patients according to the regulation of the ethical committee of Faculty of medicine Fayoum University.

Inclusion criteria:

1. Patients aged 18 to 50 years old.
2. Patient with clinically palpable varicocele with any of the following:

   * 1ry or 2ry infertility.
   * Intractable pain.
   * Affected semen parameters.
   * Reduced testicular volume.

Exclusion criteria:

1. Patients less than 18 years old.
2. Patients older than 50 years old.
3. Patients suffering from any systemic diseases that may have effect on the arterial flow like Diabetes, hypertension, liver disease and hypercholesterolemia.
4. Patients who underwent previous varicocelectomy operations or inguinoscrotal operation on the same side.
5. Sub-clinical varicocele.

   Methods:

   Preoperative assessment:

   All patients will be evaluated with full medical and surgical history stressing on:

   • Social history (special habits, marital duration, occupation, etc….)

   • Conceptional history.
   * Previous surgical procedures especially in inguinoscrotal area.
   * Sexual history. Full general and local examination, 1. physical examination: a) General and abdominal examination :
   * Age-appropriate development of male secondary sexual characteristics.
   * Gynecomastia.
   * Evaluation for lesions or scarring to the abdomen or groin. b) Local examination :
   * The scrotum must be carefully examined, and the presence of all scrotal structures should be confirmed:

     -Testicular tenderness, size, consistency and any swellings.

     - Epididymis and the Vas for nodules, presence or absence on both sides.
     * Palpating the Pampiniform plexus of the cord and grading of the varicocele in supine and standing positions, with applying Valsalva maneuver.
   * Genital examination (penis) for any abnormalities. 2. Laboratory investigations:
   * At least two semen analysis will be done to all patients before and 3 months after varicocelectomy.
   * Hormonal analysis for patients with severe oligospermia and azospermia.
   * Preoperative routine lab investigations as CBC, bleeding profile, kidney function tests and liver function tests.

     3. Radiological examination:

   Scrotal ultrasonography to asses:

   • The size and echogenicity of both testes and epididymis.

   • Peritesticular fluid collection.

   • Any abnormalities or cysts in testis or epididymis.

   Color Doppler ultrasound to assess:

   • Venous system:
   * Measurements of vein diameter.
   * Degree of reflux with Valsalva maneuver.

     • Arterial system (measurement of ):
   * Resistive index (RI) for intratesticular and capsular arteries.

     * Both U/S and Doppler will be done before and 3 months after the procedure.

   Operative technique:

<!-- -->

1. All patients will be subjected to subinguinal varicocelectomy under spinal anaesthethia / general if indicated.
2. All patients put in supine position.
3. 2-3 cm skin incision is made in a subinguinal location, just lateral to the base of the penis, a few centimeters caudal to the external ring.
4. Skin is incised sharply, and the deep dermal layer and subcutaneous adipose tissue are divided with electrocautery, taking care to stay superficial to avoid inadvertent injury to the spermatic cord.
5. Opening of Scarpa's fascia bluntly or by tip of Metzenbaum scissors.
6. Identification of the spermatic cord and its suspension above the skin.
7. Opening of the external spermatic fascia and internal spermatic fascia will expose vas deferens and vascular elements of the cord.

   In group A (Loupe-assisted group): using surgical loop (Sinirgia 3.3X Expandable field) with a magnification power of ×3.3

   • Nitroglycerin instillation on the spermatic cord using Insulin syringe drop by drop (1 cc) to help in identification and isolation of the testicular artery and more identification of affected veins.

   • Close monitoring of blood pressure by the anesthesiologist while using nitroglycerin as it may cause hypotension.

   • All abnormally dilated internal spermatic veins and external spermatic veins will be ligated with 3-0 vicryl suture with preservation of testicular artery, vasal vessels and lymphatics.

   In group B (Microscopic group): Using surgical microscope with ×10 to ×12 magnification power to identify testicular artery and lymphatics.
   * All abnormally dilated internal spermatic veins and external spermatic veins will be ligated with 3-0 vicryl suture with preservation of testicular artery, vasal vessels and lymphatics.
8. Closure of the layers of the spermatic fascia.
9. Closure of Scapa's fascia.
10. Closure of the skin with subcuticular sutures using 3-0 vicryl suture.

Intraoperative data:

* Total time of operation calculated from the start of skin incision to its closure.
* Number of ligated veins (outside the cord and inside it).
* Vital signs observation during the procedure.

Postoperative period:

All patients will be observed post operatively regarding:

• Vital signs.

• Bleeding.

* Scrotal hematoma.
* Postoperative hospital stay.

Follow up:

All patients will be followed up regularly at least for 3 months post-operative and will be evaluated with new semen analysis and new scrotal Doppler at the end of the 3 months.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 18 to 50 years old.
2. Patient with clinically palpable varicocele with any of the following:

   * 1ry or 2ry infertility.
   * Intractable pain.
   * Affected semen parameters.
   * Reduced testicular volume.

Exclusion Criteria:

1. Patients less than 18 years old.
2. Patients older than 50 years old.
3. Patients suffering from any systemic diseases that may have effect on the arterial flow like Diabetes, hypertension, liver disease and hypercholesterolemia.
4. Patients who underwent previous varicocelectomy operations or inguinoscrotal operation on the same side.
5. Sub-clinical varicocele.

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2024-05-01 (Actual); Study Completion 2024-05-01 (Actual)

PRIMARY OUTCOMES:
To assess the efficacy and safety of Loupe varicocelectomy using nitroglycerine to induce vasodilatation during operation. | 3 months follow up
  by assessing number of ligated veins, visualization of artery (during operation), and to assess PSV & EDV for testicular artery, & semen parameter (After 3 months Post operation )

SECONDARY OUTCOMES:
to assess the efficacy and safety of nitroglycerine instillation during Loupe varicocelectomy comparing to the standard Microscopic varicocelectomy. | 3 months follow up
  by assessing number of ligated veins, visualization of artery (during Loupe varicocelectomy using nitroglycerine instillation during operation), and to assess PSV & EDV for testicular artery & semen parameter (After 3 months Post operation) comparing to the standard Microscopic varicocelectomy.

CONTACTS AND LOCATIONS:
Locations (1):
- Fayoum University Hospital, Al Fayyum, Egypt